CLINICAL TRIAL: NCT04752670
Title: Prospective Registry of Submucosal Endoscopic Procedures Performed by a Novel Electrosurgical Unit
Brief Title: ConMed Beamer Study
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Principal Investigator, Mohamed Othman, M.D. Director of Advanced Endoscopy Assistant Professor of Medicine - Gastroenterology Section, Baylor College of Medicine
Other Study IDs: H-49160
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Gastrointestinal Neoplasms; Achalasia; Gastroparesis
Keywords: Endoscopic Submucosal Dissection; Per-Oral Endoscopic Myotomy (POEM); Gastric Per-Oral Endoscopic Myotomy (G-POEM)
MeSH Terms: conditions — Gastrointestinal Neoplasms; Esophageal Achalasia; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective registry of all patients who endoscopic submucosal dissection (ESD), per-oral endoscopic myotomy (POEM) and gastric per-oral endoscopic myotomy (G-POEM) using ConMed Electrosurgical unit for submucosal Dissection at Baylor St Luke's Medical Center. Collected information includes; procedure technical success rate, duration, periprocedural complications and ease of use.

DETAILED DESCRIPTION:
Submucosal endoscopy is a novel subset of procedures which enables endoscopist to utilize the submucosal space to perform advanced endoscopic procedures. The submucosa is the third layer of the gastrointestinal wall and it is a potential space which is expandable upon injecting the submucosa with fluid. The expanded submucosa causes a significant lift which enable dissection of the submucosal space with the removal of the overlying polyp or early cancer. The submucosal space can be also utilized to create a longitudinal submucosal tunnel in the esophagus or the stomach wall which allows for performing lower esophageal sphincter or pyloric myotomy for the treatment of achalasia or Gastroparesis.

Currently, the most commonly performed submucosal endoscopy procedures are endoscopic submucosal dissection (ESD) for removal of early cancers or polyps throughout the gastrointestinal tract, Per-oral Endoscopic Myotomy (POEM) for treatment of achalasia, or Gastric Per-Oral Endoscopic myotomy for the treatment of Gastroparesis. All of the above procedures require a specialized electrosurgical unit (ESU) which generate high frequency current to help incision (cutting) of the mucosa and dissection (coagulation) of the submucosa. The ConMed Beamer is a novel ESU with tissue sensing property which expedites the process of submucosal dissection. The device is currently approved for clinical use in the US. The purpose of this study is to create registry for all submucosal endoscopy procedures performed using ConMed Beamer device at BSLMC with focus on clinical outcomes of the procedure including adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old
* Patient is capable of providing informed consent
* Patient is referred for endoscopic submucosal dissection, per-oral endoscopic myotomy, or gastric per-oral endoscopic myotomy

Exclusion Criteria:

* Patient is < 18 years old
* Patient refused and/or unable to provide consent
* Patient is a pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for an ESD, POEM or GPOEM satisfying all eligibility criteria will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Technical Success rate | 1 year
  Defined as the ability to perform the entire procedure using the ConMed Beamer electrosurgical system

SECONDARY OUTCOMES:
Procedure Time | 1 year
  Determine length of time to perform procedure using ConMed Beamer electrosurgical system
Adverse Events | 1 year
  Intraprocedural AE such as bleeding or perforation
Adverse Events | 1 year
  Post procedural, post polypectomy, delayed bleeding or delayed perforation

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor St. Lukes Medical Center (BSLMC), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a prospective single-center registry study.